CLINICAL TRIAL: NCT03220022
Title: A Pilot Study of Ibrutinib and R-da-EPOCH for Front Line Treatment of AIDS-Related Lymphomas
Brief Title: Ibrutinib, Rituximab, Etoposide, Prednisone, Vincristine Sulfate, Cyclophosphamide, and Doxorubicin Hydrochloride in Treating Patients With HIV-Positive Stage II-IV Diffuse Large B-Cell Lymphomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01240; NCI-2017-01240 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-101 (Other: AIDS Malignancy Consortium); AMC-101 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: AIDS-Related Lymphoma; Ann Arbor Stage II Diffuse Large B-Cell Lymphoma; Ann Arbor Stage III Diffuse Large B-Cell Lymphoma; Ann Arbor Stage IV Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, AIDS-Related | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; ibrutinib; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (R-da-EPOCH) (Experimental): Patients receive rituximab IV on day 1 (for CD20 positive patients only), etoposide IV over 96 hours on days 1-4, doxorubicin hydrochloride IV over 96 hours on days 1-4, vincristine sulfate IV over 96 hours on days 1-4, prednisone PO daily on days 1-5, cyclophosphamide IV over 1 hour on day 5, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive pegfilgrastim SC from 1 calendar day up to 48 hours or filgrastim SC beginning on day 6 for up to 10 days until ANC is satisfactory.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Pegfilgrastim; Other: Pharmacological Study; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase I trial studies the side effect and best dose of ibrutinib in combination with rituximab, etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride in treating patients with human immunodeficiency virus (HIV)-positive stage II-IV diffuse large B-cell lymphomas. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib and etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride may work better in treating patients with HIV-positive diffuse large B-cell lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of ibrutinib and rituximab (R)-dose adjusted (da)-etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride (EPOCH) in participants with acquired immunodeficiency syndrome (AIDS)-related lymphomas (ARL).

SECONDARY OBJECTIVES:

I. To evaluate the complete response (CR) rates of ARL to ibrutinib and R-da-EPOCH.

II. To measure the 1-year and 2-year overall and progression-free survival of participants with ARL treated with combination ibrutinib and R-da-EPOCH, including preliminary comparison of non-germinal center B-cell (GCB) with historical controls treated with R-da-EPOCH.

III. To categorize and compare the cell-of-origin by gene expression profiling (GEP) gene expression-based classification (GCB, activated B-cell-like, unclassifiable) to immunohistochemistry (IHC) classification (GCB, non-GCB), estimate the discordant classification, and correlate each biological classification (IHC and GEP) with treatment response rates and survival.

IV. To calculate the percentage of participants who receive two or more cycles of R-da-EPOCH, and are able to continue on a minimum dose level of cyclophosphamide of -1 and above after dose adjustments for hematologic toxicities.

V. To determine the average number of days per cycle participants are able to stay on planned dose of ibrutinib at the recommended phase II dose (RP2D).

VI. To assess the effect of ibrutinib and R-da-EPOCH on levels of circulating tumor deoxyribonucleic acid (DNA).

VII. To assess the effect and degree of ibrutinib and R-da-EPOCH on T-cell receptor signaling via ITK inhibition.

VIII. To assess the effect of ibrutinib and R-da-EPOCH on B-cell receptor signaling pathway including BTK activity in ARL.

IX. To evaluate the soluble cytokine response to ibrutinib and R-da-EPOCH. X. To characterize the pharmacokinetics of doxorubicin, etoposide, and vincristine in the presence of ibrutinib, and vice versa, and assess the clinical relevance of any drug-drug interaction and correlate with pharmacodynamics outcomes.

OUTLINE: This is a dose escalation study of ibrutinib.

Patients receive rituximab intravenously (IV) on day 1 (for CD20 positive patients only), etoposide IV over 96 hours on days 1-4, doxorubicin hydrochloride IV over 96 hours on days 1-4, vincristine sulfate IV over 96 hours on days 1-4, prednisone orally (PO) daily on days 1-5, cyclophosphamide IV over 1 hour on day 5, and ibrutinib PO once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive pegfilgrastim subcutaneously (SC) from 1 calendar day up to 48 hours or filgrastim SC beginning on day 6 for up to 10 days until absolute neutrophil count (ANC) is satisfactory.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically (via at least a core or ideally, incisional or excisional biopsy) documented CD20 positive or negative diffuse large B-cell lymphoma (DLBCL)
* Tissue available from the diagnostic biopsy in the form of blocks, tissue cores, or slides available for submission to central pathology is required for all participants enrolled to this study, for analysis of integral biomarkers. Formalin-fixed paraffin-embedded tissue from diagnostic tissue is acceptable and recommended; submission of the institutional diagnostic slides is also preferred for all participants enrolled in the study. Tissue and diagnostic slides are required to be submitted within 1 month of enrollment
* Stage II-IV disease; participant will need measurable disease by computed tomography (CT) or positron emission tomography (PET) scans if enrolled in the dose-expansion cohort
* HIV positive; documentation of HIV-1 infection by means of any one of the following:

  * Documentation of HIV diagnosis in the medical record by a licensed health care provider;
  * Documentation of receipt of ART (at least three different medications) by a licensed health care provider (documentation may be a record of an antiretroviral therapy (ART) prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name);
  * HIV-1 ribonucleic acid (RNA) detection by a licensed HIV-1 RNA assay demonstrating > 1000 RNA copies/mL;
  * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 western blot confirmation or HIV rapid multispot antibody differentiation assay
  * NOTE: a "licensed" assay refers to a United States (U.S.) Food and Drug Administration (FDA)-approved assay, which is required for all investigational food drug (IND) studies
* For the dose-finding cohort participants lymphoma must be untreated. For the dose-expansion cohort participants may have either untreated lymphoma or may have received prior therapy
* Ages 18 - 64
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* For the dose-finding cohort participants must have a CD4 count ≥ 100 cells/mm^3. For the dose-expansion cohort participants may have any CD4 count, including a CD4 count < 100 cells/mm^3
* Absolute neutrophil count: >= 1,000/mm^3, unless decreased due to bone marrow involvement with lymphoma
* Platelets: >= 75,000/mm^3, unless decreased due to bone marrow involvement with lymphoma
* Total bilirubin: =< 1.5 times the institutional upper limit of normal (ULN); if potentially due to lymphoma, in the dose-expansion cohort, the first cycle may be given without ibrutinib and if transaminitis and bilirubinemia improves to meet parameters, participant may be enrolled
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): < 2 times the institutional ULN; if potentially due to lymphoma, in the dose-expansion cohort, the first cycle will be given without ibrutinib and if transaminitis and bilirubinemia improves to meet parameters, participant may be enrolled
* Creatinine levels below the normal institutional upper limits; or, creatinine clearance >= 50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal; unless decreased due to renal involvement by lymphoma
* Participants must not be on medications, including antiretroviral (ARV) regimens such as cobicistat, indinavir, or ritonavir, or agents with moderate or strong CYP3A4 inhibition; if on a moderate or strong CYP3A4 inhibitor regimen prior to study enrollment, participants must be switched to a qualifying regimen with the last dose of the strong CYP3A4 inhibitor taken at least one week before administration of ibrutinib
* Willingness of sexually active participants to use adequate contraception; both men and women of child-bearing potential treated or enrolled on this study must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before study entry, for the duration of study participation, 90 days after completion of ibrutinib, and 12 months after the last dose of rituximab, whichever comes last; men who only have sex with other men do not need to use contraception specifically for this study (should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately)
* All participants will be required to be screened for hepatitis B; all participants who present with acute hepatitis B or show normal transaminases and are hepatitis B surface antigen (HBsAg) positive (+) and IgM+ for hepatitis core antigen will not be eligible for trial enrollment; per Infectious Diseases Society of America (IDSA) and Assistance for AIDS Specific Drugs (AASD) guidelines, those participants that show no immunity, defined by the lack of hepatitis B surface antibody, and show evidence of chronic infection (i.e. hepatitis B [HB]sAg+, HBcore+, hepatitis B surface antibody [HBsAB] negative [-]) will be required to be on anti-hepatitis B therapy, during the study, in order to be eligible; the exact hepatitis B therapy will be at the discretion of the infection disease specialist or investigator; if infected with hepatitis B, participants will be permitted to enroll in the study provided liver function tests meet criteria listed above, there is no evidence of cirrhosis AND participants will be required to be on anti-hepatitis B therapy
* All participants will be required to be screened for hepatitis C; if hepatitis C antibody positive, with or without a positive hepatitis C RNA level, participants will be permitted to enroll in the study provided liver function tests meet criteria listed, and have no evidence of cirrhosis; participants diagnosed with hepatitis C less than 6 months from trial enrollment will be considered to have acute hepatitis C, and will be excluded from study UNLESS hepatitis C viral load is undetectable
* Adequate cardiac function defined as an ejection fraction on echocardiogram (ECHO) or multi-gated acquisition (MUGA) that is at or above the institutional normal limits. For the dose-expansion cohort, if the participant had a pre-treatment ECHO prior to pre-study therapy which reports adequate cardiac function defined as an ejection fraction on ECHO or MUGA that is at or above the institutional normal limits, a repeat ECHO will not need to be repeated prior to start of study treatment
* Participants must be able to swallow oral pills
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy other than R-EPOCH, R-CHOP, or limited therapy, or radiotherapy other than palliative radiation for medical emergencies (like cord compression), within the last 4 weeks
* For the dose-finding cohort prior cytotoxic chemotherapy or radiotherapy for this lymphoma is exclusionary. For the dose-expansion cohort participants may have received:

  * A maximum of one cycle of combination chemotherapy, including rituximab-containing regimens R-CHOP and R-EPOCH. The start of previous chemotherapy cycle must occur at least 21 days but no more than 28 days prior to beginning treatment under this protocol, and such cycle will count towards the maximum of 6 cycles under this study (i.e., cycle off study will count as cycle 1) OR
  * 1 prior cycle of limited therapy including cyclophosphamide and/or rituximab and/or glucocorticoids to improve hepatic or renal function impaired due to lymphoma involvement. The start of this therapy may occur up to 28 days prior to beginning treatment under this protocol; cyclophosphamide administration must have been completed at least 14 days prior to initiation of protocol therapy. Such treatment will not count towards the maximum of 6 cycles under this study (i.e., participants will receive 6 cycles on study)
* For the dose-finding cohort rituximab within 12 months prior to study registration will be exclusionary; only exception will be if rituximab was given for indications other than the treatment of aggressive lymphoma. For the dose-expansion cohort one cycle of rituximab as part of R-CHOP or R-EPOCH or limited therapy may be administered off study prior to enrollment; prior rituximab will also be allowed if rituximab was given for indications other than the treatment of aggressive lymphoma
* Participants who are receiving any other investigational agents
* Participants who have previously received ibrutinib for another indication
* Expected survival < 2 months
* Participants with a history of an opportunistic fungal infection or active fungal infection requiring, or at high risk of requiring, prophylactic or treatment with fluconazole, voriconazole or posaconazole
* Participants with known brain metastases from solid tumors should be excluded from this clinical trial
* Presence of second active tumor, other than non-melanoma skin cancer, carcinoma in situ of the cervix, or Kaposi's sarcoma (KS) that requires systemic therapy
* For the dose-finding cohort, participants with known or suspected parenchymal brain, spinal cord, leptomeningeal disease prior to study enrollment will be excluded. For the dose-expansion cohort participants with known or suspected parenchymal brain or spinal cord disease, or symptomatic leptomeningeal disease will be excluded. Asymptomatic leptomeningeal disease will be allowed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinions of the investigator, would limit compliance with study requirements
* Pregnancy or breastfeeding; a pregnancy test must be performed within 7 days prior to ibrutinib initiation in women of childbearing potential; pregnant women; breastfeeding must be discontinued because of unknown but potential risks in the nursing infant
* Unable to comply with the requirements of the protocol, or unable to provide adequate informed consent in the opinion of the principal investigator
* Serious, ongoing, non-malignant disease or infection, which in the opinion of the investigator and/or the sponsor would compromise other protocol objectives; participants with active opportunistic infections are ineligible
* Major surgery, other than diagnostic surgery, occurring 4 weeks prior to study entry; splenectomy will not be considered an exclusionary major surgery
* History of cutaneous or mucocutaneous reactions, or diseases in the past, due to any cause, severe enough to cause hospitalization or an inability to eat or drink for > 2 days; this exclusion relates to the long-term possibility of severe cutaneous or mucocutaneous reactions to rituximab that might occur at increased frequency in participants who have had severe skin disease or reactions in the past
* Myocardial infarction (MI) within 6 months prior to study entry, New York Heart Association (NYHA) class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ibrutinib in combination with chemotherapy | Up to 21 days
  Will be descriptive and will be reported in tabular format with the appropriate summary statistics (count and percentage). In the dose-finding portion, the number of dose limiting toxicities (DLTs) identified among the DLT-evaluable subjects will be listed and summarized by dose level. The safety variables will be listed and summarized for (1) subjects in the dose-finding portion, (2) subjects in the dose expansion cohort (DEC), and (3) all subjects in the study.
Recommended phase II dose (RP2D) of ibrutinib in combination with chemotherapy | Up to 21 days
  Will be descriptive and will be reported in tabular format with the appropriate summary statistics (count and percentage). In the dose-finding portion, the number of DLTs identified among the DLT-evaluable subjects will be listed and summarized by dose level. The safety variables will be listed and summarized for (1) subjects in the dose-finding portion, (2) subjects in the DEC, and (3) all subjects in the study.

SECONDARY OUTCOMES:
Incidence of adverse events graded using Common Terminology Criteria for Adverse Events version 4.0 | Up to 5 years
  Toxicity data will be presented by type and severity for each dose cohort. Incidence of toxicity related dose reductions and treatment discontinuations will be summarized for each dose group.
Complete response rates | Up to 5 years
  The complete response rates and their corresponding 95% confidence intervals will be calculated for participants with AIDS-related lymphomas (ARL) treated with combination ibrutinib and rituximab (R)-dose adjusted (da)-etoposide, prednisone, vincristine sulfate, cyclophosphamide and doxorubicin hydrochloride (EPOCH).
Progression free survival (PFS) | 1 year
  PFS will be estimated using Kaplan Meier method, as well as, their corresponding 95% confidence intervals.
Progression free survival (PFS) | 2 years
  PFS will be estimated using Kaplan Meier method, as well as, their corresponding 95% confidence intervals.
Overall survival (OS) | 1 year
  OS will be estimated using Kaplan Meier method, as well as, their corresponding 95% confidence intervals.
Overall survival (OS) | 2 years
  OS will be estimated using Kaplan Meier method, as well as, their corresponding 95% confidence intervals.
Lymphoma cell-of-origin (COO) assessment | Up to 5 years
  Will be determined by gene expression profiling (GEP) (germinal center B-cell [GCB], activated B-cell [ABC], unclassifiable) and immunohistochemistry [IHC] (GCB, non-GCB). The concordances and discordances between classifications will be estimated with binomial proportions and their 95% corresponding confidence intervals. The response rates and survival as categorized by GEP or IHC will be compared, to see which analysis of COO best correlates with treatment response. Chi-square tests will be used to test the associations between 1) GEP (GCB, ABC, unclassifiable) with response rates and 2) IHC (GCB, non-GCB) with responses rate. The Kaplan Meier method will be used to calculate estimates of OS and PFS within GEP (GCB, ABC, unclassifiable) and within IHC (GCB, non-GCB), as well as their 95% confidence intervals. The log-rank test will be used to test differences with respect to OS and PFS within GEP and within IHC.
Percentage of participants who receive two or more cycles of combination chemotherapy, and are able to continue on a minimum dose level of cyclophosphamide of -1 and above after dose adjustments | Up to 5 years
  Hematologic toxicities will be calculated.
Average number of days per cycle participants are able to stay on planned dose of ibrutinib | Up to 5 years
  Average number of days will be calculated.
Changes in the levels of human immunodeficiency virus (HIV)-1 viral reservoirs | Baseline up to 5 years
  Descriptive statistics will be used to evaluate the changes and will be compared with treatment completion. If there are sufficient data, the binomial test of proportions will be used to test if the long term viral reservoir is either undetectable or below baseline in at least half of the participants.
Changes in Epstein-Barr virus (EBV) viral loads | Baseline up to 5 years
  Descriptive statistics will be used to evaluate the changes and compared with treatment completion. If there are sufficient data, the binomial test of proportions will be used to test if the long term viral reservoir is either undetectable or below baseline in at least half of the participants.
Effect of treatment on HIV latency reservoirs | Up to 5 years
  Will be correlated with degree of ITK inhibition and Pearson or Spearman correlation coefficients will be used, as appropriate.
Effect of treatment on B-cell receptor signaling pathway including BTK activity | Up to 5 years
  Descriptive statistics will be used.
Effect of treatment on T-cell receptor signaling via ITK activity. | Up to 5 years
  Descriptive statistics will be used.
Soluble cytokine response to treatment | Up to 5 years
  Descriptive statistics will be used.
Pharmacokinetics (PK) parameters assessment for ibrutinib, doxorubicin hydrochloride, etoposide, and vincristine sulfate | Up to 5 years
  Relevant individual PK parameters will be estimated using non-compartmental or compartmental PK methods with the software WinNonlin. The PK variables will be tabulated and descriptive statistics (e.g., geometric means and coefficients of variation) and compared across dose levels (if applicable) using nonparametric statistical testing techniques. PK parameters (i.e., steady state concentration [Css], clearance [Cl], and area under the curve [AUC]) will be correlated with pharmacodynamics effects using nonparametric statistical testing techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Ida C Wong-Sefidan, Principal Investigator — AIDS Malignancy Consortium
Locations (19):
- United States (19):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois College of Medicine - Chicago, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington